CLINICAL TRIAL: NCT07322068
Title: Perennial Malaria Chemoprevention in the Malaria Vaccine Era
Acronym: PMC-VAC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); Infectious Diseases Research Collaboration, Uganda (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Prasanna Jagannathan, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 84540
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PMC-Placebo (Placebo Comparator): Placebo given at Expanded Program of Immunization (EPI) visits (8 doses of placebo at 2.5, 3.5, 6, 7, 8, 9, 12, and 18 months of age).
  Participants will receive DP placebo plus SPAQ placebo. Placebos with an identical appearance to either DP or SPAQ active drugs will be provided by their manufacturers.
  Interventions: Drug: Dihydroartemisinin Piperaquine Placebo; Drug: Sulfadoxine pyrimethamine + Amodiaquine placebo
- PMC-SPAQ (Experimental): Perennial malaria chemoprevention with sulfadoxine-pyrimethamine + amodiaquine (SPAQ) given at Expanded Program of Immunization (EPI) visits (8 doses of SPAQ at 2.5, 3.5, 6, 7, 8, 9, 12, and 18 months of age).
  Participants will also receive DP placebo along with active SPAQ. Placebo with an identical appearance to DP active drug will be provided by its manufacturer.
  Interventions: Drug: Sulfadoxine pyrimethamine + Amodiaquine; Drug: Dihydroartemisinin Piperaquine Placebo
- PMC-DP (Experimental): Perennial malaria chemoprevention with dihydroartemisinin-piperaquine (DP) given at Expanded Program of Immunization (EPI) visits (8 doses of DP at 2.5, 3.5, 6, 7, 8, 9, 12, and 18 months of age).
  Participants will also receive SPAQ placebo along with active DP. Placebo with an identical appearance to SPAQ active drug will be provided by its manufacturer.
  Interventions: Drug: Dihydroartemisinin Piperaquine; Drug: Sulfadoxine pyrimethamine + Amodiaquine placebo

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine + Amodiaquine — Each round of study drugs will consist of once daily oral dosing x 3 days. The first daily dose will be directly observed in the study clinic, and day 2 and day 3 doses will be provided for administration at home. Daily dosing of SPAQ will be based on manufacturer's recommendations: infants <12 months of age will receive one dose of 12.5/250 mg SP and 3 daily doses of 76.5 mg AQ, children >=12 months of age will receive one does of 25/5000 mg SP and 3 daily doses of 153 mg AQ.
  Other Names: SPAQ
  Arms: PMC-SPAQ
Drug: Dihydroartemisinin Piperaquine — Each round of study drugs will consist of once daily oral dosing x 3 days. The first daily dose will be directly observed in the study clinic, and day 2 and day 3 doses will be provided for administration at home. Daily dosing of DP will consist of half-strength tablets given once a day for 3 consecutive days and will depend on bodyweight, targeting 4 mg/kg of dihydroartemisinin and 24 mg/kg of piperaquine phosphate.
  Other Names: DP
  Arms: PMC-DP
Drug: Dihydroartemisinin Piperaquine Placebo — Participants receive oral placebos with an identical appearance to DP active drug.
  Other Names: DP Placebo
  Arms: PMC-Placebo; PMC-SPAQ
Drug: Sulfadoxine pyrimethamine + Amodiaquine placebo — Participants receive oral placebos with an identical appearance to SPAQ active drug.
  Other Names: SPAQ Placebo
  Arms: PMC-DP; PMC-Placebo

SUMMARY:
Malaria remains a major cause of pediatric deaths and morbidity in Africa. An affordable malaria vaccine, R21, is being deployed in Uganda and other African countries with high malaria transmission, but efficacy is incomplete and wanes rapidly, and R21 does not provide protection until infants complete the primary vaccination series, or ~9 months of age. The goal of this study is to see whether combining R21 vaccination with two novel perennial malaria chemoprevention regimens can enhance protection against malaria compared with R21 alone. This study will take place at Masafu General Hospital (MGH) in Busia District, a rural area in Southeastern Uganda bordering Lake Victoria.

ELIGIBILITY:
Inclusion Criteria:

* Residency in Busia District, Uganda
* Provision of informed consent by the parent/guardian for her child
* Agreement to come to the study clinic for any febrile episode or other illness and avoid, where possible, medications given outside the study protocol

Exclusion Criteria:

* Intention of permanently moving outside Busia district during the study period
* Active medical problem requiring inpatient evaluation or chronic medical condition requiring frequent medical attention at the time of screening
* Evidence of sickle cell disease (Hemoglobin SS genotype)
* Biological mother known to be HIV positive

Ages: 1 Day to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1290 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic malaria | 2.5 months to 60 months of age
  The incidence of symptomatic malaria is defined as the number of incident episodes of malaria requiring treatment per time at risk. Treatments within 14 days of a prior episode are not considered incident events.

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Jagannathan, MD, Principal Investigator — Stanford University
Locations (1):
- Masafu General Hospital, Busia District, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Clinical data will be recorded on case report forms, a study database will be updated monthly, and available (blinded) data will be shared with project investigators. Monthly reports will be generated for all investigators, including data summaries, number and type of assays performed, quality control checks, etc. To facilitate interpretation of the data, study protocols, data dictionaries, and documentation related to any of the data described above will be made publicly available. The same is true for any additional metadata used in the analyses resulting in publications including data on interventions. For parasite genomic and host immunologic data deposited in public repositories (e.g. GEO, IMMPORT), project, study, sample, experimental, and file level metadata will be provided using templates provided by GEO and SRA data repositories or IMMPORT.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All scientific data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first.